CLINICAL TRIAL: NCT00133458
Title: Randomized, Double Blind Comparison of Two Lenghts of Albendazole Therapy for Subarachnoid Cysticercosis
Brief Title: RCT ALB for SA Cysticercosis
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 04-003
Record Dates: First submitted 2005-08-19; First posted 2005-08-23 (Estimated); Last update posted 2019-01-30 (Actual); Status verified 2005-10

CONDITIONS: Subarachnoid Cysticercosis
Keywords: Albenza, Subarachnoid cysticercosis
MeSH Terms: interventions — Albendazole

INTERVENTIONS:
Drug: Albendazole

SUMMARY:
This study will enroll 120 individuals diagnosed with subarachnoid cysticercosis, a disease caused by the invasion of the basal part of your brain by a parasite named Taenia solium. Subarachnoid cysticercosis is usually treated with albendazole for one month to kill the parasite. This study will determine if two months of albendazole (ABZ) therapy is better than one-month. The study will last 3 years.

DETAILED DESCRIPTION:
This is a randomized, double blind comparison of two lengths of albendazole thereapy for subarachnoid cysticercosis. It will enroll 120 individuals, male and female age 18 to 65, and diagnosed with subarachnoid cysticercosis, a disease caused by the invasion of the basal part of your brain by a parasite named Taenia solium. Subarachnoid cysticercosis is usually treated with albendazole for one month to kill the parasite. This study will determine if two months of albendazole (ABZ) therapy is better than one-month. The study will last 3 years.

ELIGIBILITY:
Inclusion Criteria:

* Male or female individuals between 18-65 year of age with a diagnosis of basal subarachnoid cysticercosis, based on MRI and confirmed by serological test.
* Willingness to accomplish the two weeks minimal hospitalization required.
* Female of child-bearing potential willing to use an adequate method of contraception including implants, injectables, combined oral contraceptives, effective intrauterine devices, sexual abstinence, or vasectomized partner while participating in the study.
* Patients with normal laboratory values for hemoglobin, platelet counts, total white blood cells, glucose, creatinine, bilirubin, ALT, AST, and electrolytes.
* Negative fecal exam for Taenia eggs.

Exclusion Criteria:

* Previous therapy with albendazole (does not include patients who received single-dose 400 mg ABZ for intestinal parasites), or praziquantel.
* Pulmonary tuberculosis evidenced by a positive chest X-ray and positive sputum smears.
* Pre-existing diagnosis of diabetes
* Systemic disease other than NCC that may affect therapy or short-term prognosis, including but not limited to chronic renal failure, hepatic insufficiency, cardiac failure, and steroid-dependent immune diseases. Identification of systemic diseases will be left to the discretion of each Site PI.
* Patients in unstable condition or with severe intracranial hypertension (ICH). Definition of severe ICH for this study would be the presence of headaches, nausea, and vomiting and papilledema at fundoscopic examination (all of them). Patients in this category can be considered for entrance into the study only after treatment of ICH by ventricle-peritoneal shunting. Patients with CT findings compatible with intracranial hypertension will have neurosurgical evaluation (by non study personal) before study entry.
* Pregnancy
* History of hypersensitivity to albendazole
* Concurrent treatment with praziquantel, cimetidine or teophylline.
* Chronic alcohol or drug abuse

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Study Completion 2007-06

CONTACTS AND LOCATIONS:
Locations (4):
- Facultad de Medicina de Riberao, Riberao Preto, Brazil
- Instituto Neurologico de Antioquia, Medellín, Colombia
- Neurology Service, Hospital -Clinica Kennedy, Guayaquil, Ecuador
- Universidad Peruana Cayetano Heredia, Lima, Peru